CLINICAL TRIAL: NCT01862939
Title: A Double Blind, Placebo-Controlled, Randomized, Two-Part, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of DS-7309 in Healthy Volunteers and Subjects With Type 2 Diabetes Mellitus
Brief Title: A Two-Part, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of DS-7309 in Healthy Volunteers and Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: DS7309-A-U101
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- part 1 DS-7309 ascending dose (Experimental): 1, 2.5, 5, 10, 20 mg blinded DS-7309 powder in bottle.
  Interventions: Drug: DS-7309
- part 2 DS-7309 (Experimental): 1, 2.5, 5, and 15mg DS-7309 powder in bottle for oral solution.
  Interventions: Drug: DS-7309
- part 2 placebo (Placebo Comparator): placebo to match part 2 DS-7309
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: DS-7309 — 1, 2.5, 5, 10, 20 mg DS-7309 powder in bottle.
  Arms: part 1 DS-7309 ascending dose; part 2 DS-7309
Drug: placebo — placebo to match part 2 DS-7309
  Arms: part 2 placebo

SUMMARY:
This is a randomized, placebo-controlled, 2-part, sequential, single ascending dose study.

Part 1 is planned as 6 sequential escalation treatment groups. Part 2 is a randomized, placebo-controlled, two-period sequential pharmacodynamic (PD) arm.

ELIGIBILITY:
Inclusion Criteria:

* Women must be of non-child bearing potential, ie, either:

  1. Surgically sterile (ie, bilateral tubal ligation or removal of both ovaries and/or uterus at least 6 months prior to dosing), or
  2. Naturally postmenopausal (spontaneous cessation of menses) for at least 24 consecutive months prior to dosing, with a follicle stimulating hormone (FSH) level at screening of ≥ 40 mIU/mL.
* All women must have a negative serum pregnancy test at screening and within 48 hours before dosing.
* Able to understand and willing to comply with all study requirements, and willing to follow the study medication regimen.
* Subjects must give written informed consent to participation in the study prior to screening.
* Negative urine test for drugs of abuse and alcohol at screening and check-in.
* Negative result for HIV antibody, hepatitis B surface antigen, and hepatitis C antibody at screening.
* Subjects must agree to abstain from alcohol, cola, tea, coffee, chocolate and other caffeinated drink and food from 2 days before check-in and throughout confinement.
* Subjects must agree to abstain from grapefruit/grapefruit juice and Seville oranges from 10 days before the first dose and throughout the study.
* Healthy women who are not of childbearing potential and men, 18 to 45 years of age, inclusive.
* Body Mass Index (BMI) of 19.00 to 32.00 kg/m2 inclusive.
* Good health, as determined by the absence of clinically significant deviation from normal, based on medical history, physical examination, laboratory reports, and 12-lead ECG, as deemed by the Investigator, prior to enrollment.
* Baseline (0 hour) pre-dose capillary blood glucose ≥ 70 mg/dL. Part 2 (T2DM subjects)
* Women who are not of childbearing potential and men, 18 to 55 years of age, inclusive.
* Diagnosis of type 2 diabetes mellitus for a minimum of 3 months prior to first dose.
* Body Mass Index (BMI) of 19.00 to 40.00 kg/m2 inclusive.
* Subjects should be either:

  1. Treatment naïve from any antidiabetic treatment for at least 6 months prior to screening with a hemoglobin A1c (HBA1c) value between 7%-10%, inclusive.
  2. On metformin alone with a HBA1c value between 7%-9%, inclusive, and willing to discontinue current metformin treatment for at least 2 weeks prior to study and during the duration of the study. See Section 9.10.1 for monitoring during 2 week washout.

Exclusion Criteria:

* Female subject is of childbearing potential, is pregnant (as based on test results) or is breast feeding.
* Male subjects should ensure use of condom and spermicide from dosing until 12 weeks after dosing.
* Male subjects must agree not to donate sperm from dosing until 12 weeks after dosing.
* Any history of drug abuse.
* History of alcohol addiction during the 2 years prior to Day 1.
* History or current evidence, as determined by the Investigator, of psychiatric or emotional problems which would invalidate giving informed consent or limit the ability of the subject to comply with study requirements.
* History or current alcoholic or non-alcoholic liver disease or liver steatosis.
* History of neuropathy.
* Subjects with QTcF interval duration >450 msec obtained from the ECG taken at screening, after at least 10 minutes of quiet rest in a supine position.
* Subjects with a family history of long QT syndrome.
* Subjects with any history of arrhythmia.
* Significant blood donation or significant blood loss within the 56 days before Day -1.
* Plasma donation within 7 days before Day -1.
* Participation in another investigational new drug research study within the 30 days before Day 1.
* Use of tobacco products or nicotine-containing products (including smoking cessation aids, such as gums or patches) within the 6 months before Day 1.
* Relationship of the subject to the Investigator, any sub-investigator, pharmacist, study coordinator, or other staff directly involved in the conduct of the study, or employment by the Sponsor or contract research organization participating in the study.
* Familial relationship of the subject to any subjects previously or currently enrolled in the study.
* Screening laboratory values outside the range of normal values that are deemed clinically significant by the Investigator. Liver function tests (AST, ALT, total bilirubin, and lactate dehydrogenase [LDH]) must be at or below the ULN. If a subject has a non-clinically significant high abnormal reading for one or more of the liver function tests on the screening lab test, the test may be repeated once. If the lab test results are normal on the repeat test, he/she may be enrolled provided the Day -1 lab test results are also normal.
* Hemoglobin levels below the lower limit of normal of the clinical laboratory's reference range at the screening visit.
* Enrollment in a prior dose cohort of this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
incremental area under the curve (IAUC) blood glucose | 5 hours
  The incremental area under the curve (IAUC) of the PD biomarker blood glucose following an oral glucose tolerance test (OGTT) in subjects with type 2 diabetes mellitus (T2DM).

SECONDARY OUTCOMES:
determine blood concentrations of DS-7309 | 48 hours
  The plasma pharmacokinetic (PK) parameters of A203-5319 (the free form of DS-7309) and relevant metabolite of DS-7309 in healthy subjects and subjects with T2DM.

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Tempe, Arizona, United States